CLINICAL TRIAL: NCT04011852
Title: The Role of Chest Electrical Impedance Tomography in the Pediatric Ventilator Weaning
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 10055719.0.0000.0068
Record Dates: First submitted 2019-07-03; First posted 2019-07-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Ventilator Weaning; Child; Spontaneous Breathing Trial; Electrical Impedance Tomography
Keywords: Ventilator Weaning; Child; Electrical Impedance Tomography; Respiration, artificial; Intensive Care units
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Electrical Impedance tomography — Monitoring with Electrical impedance tomography during spontaneous breathing trials on T-piece in children

SUMMARY:
To correlate the data obtained by Electrical impedance tomography (EIT) during the spontaneous breathing trials (SBT) on a T-piece, in children, with failure in the trial and Extubation failure.

Observe if the EIT monitoring will be able to detect the children that will fail earlier than the SBT performed alone.

Method: A cross-sectional, prospective study to explore the potential benefits of monitoring with EIT during weaning.

DETAILED DESCRIPTION:
Early and successful Extubation is sometimes a difficult combination in children, since the criteria for suggesting it are often subjective and poorly defined. Electrical impedance tomography (EIT) has been developed and used clinically for more than 30 years. Interest in this technology arose from the need to monitor ventilation and pulmonary perfusion at the bedside. Because it is a non-invasive and non-radiation technology, EIT is very promising in the pediatric population. Objectives: To correlate the data obtained by the EIT during the spontaneous breathing trials (SBT) on a T-piece with failure in the trial and Extubation failure and to observe if the EIT is able to detect the children that will fail earlier than the SBT performed alone. Method: A cross-sectional, prospective study to explore the potential benefits of monitoring with EIT during weaning. Qualitative characteristics will be described using absolute and relative frequencies and the quantitative characteristics will be described using summary measures (mean, standard deviation, median, minimum and maximum). Bivariate and later multiple logistic regression analyzes will be performed to evaluate the influence of characteristics assessed on weaning failure, mainly the reduction in functional residual capacity during and after the weaning trial. For the analysis will be used the software IBM-SPSS for Windows version 20.0 and tabulation of the data will be used Microsoft Excel 2010 software. The tests will be performed with significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

Children who are on mechanical ventilation for a period of more than 24 hours, between 28 days of age and 15 years, who are admitted to the pediatric intensive care unit (ICU) of the Children's Institute in Brazil

Exclusion Criteria:

* Upper Airway Obstruction
* Diaphragmatic hernia or diaphragmatic paralysis
* Chronic use of mechanical ventilation
* Cyanogenic congenital heart disease
* Primary pulmonary hypertension
* Neuromuscular disease
* Tracheostomy

Ages: 28 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children who are on mechanical ventilation for a period of more than 24 hours, between 28 days of age and 15 years, who are admitted to the pediatric intensive care unit (ICU) of the Children's Institute in Brazil and are ready for a weaning trial.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Correlate Electrical impedance tomography to Extubation failure | 48 hours
  Compare data obtained by the EIT during the spontaneous breathing trial with Extubation failure
Correlate Electrical impedance tomography to spontaneous breathing trial failure | 1 hour
  Observe if Electrical impedance tomography detects children who will fail in spontaneous breathing trial (during a 1-hour T-piece) earlier than clinical criteria

SECONDARY OUTCOMES:
Electrical impedance tomography Security | 2 hours
  Evaluate Electrical impedance tomography Security (skin lesion or pain)
  Neonatal Skin Condition Score
  Dryness
  1. Normal, no sign of dry skin
  2. Dry skin, visible scaling
  3. Very dry skin, cracking/fissures
  Erythema
  1. No evidence of erythema
  2. Visible erythema, < 50% body surface
  3. Visible erythema, ≥ 50% body surface
  Breakdown
  1. None evident
  2. Small, localized areas
  3. Extensive
  Note:
  Perfect score = 3 Worst score = 9
Compare tidal volume and RR / VT index with Z-delta and RR / Z-delta | 1 hour
  Verify whether traditional measures of tidal volume and the RR / VT index can be independently and accurately assessed through the measurement of Z-delta and RR / Z-delta, through the Electrical impedance tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Flávia K Foronda, MDPhD, Principal Investigator — Full staff
Locations (1):
- University of São Paulo General Hospital, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided